CLINICAL TRIAL: NCT06103266
Title: Rivaroxaban Monotherapy After CYP2C19 Genotype Testing in Patients With Atrial Fibrillation and Percutaneous Coronary Intervention
Acronym: IMPACT AF-PCI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: J.P.S Henriques (Other)
Responsible Party: Sponsor-Investigator, J.P.S Henriques, Professor doctor, Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Atrial Fibrillation; Coronary Artery Disease
MeSH Terms: conditions — Atrial Fibrillation; Coronary Artery Disease | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rivaroxaban monotherapy (Experimental): Once daily rivaroxaban 20 mg or 15 mg with reduced kidney function (eGFR 15 - 49 mmol/L) for 6 months in case of percutaneous coronary intervention for stable coronary artery disease or 12 months in case of percutaneous coronary intervention for acute coronary syndrome without concurrent antiplatelet therapy
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Rivaroxaban — Once daily rivaroxaban 20 mg or 15 mg with reduced kidney function (eGFR 15 - 49 mmol/L) for 6 months in case of percutaneous coronary intervention for stable coronary artery disease or 12 months in case of percutaneous coronary intervention for acute coronary syndrome without concurrent antiplatelet therapy

SUMMARY:
Rationale: Patients with atrial fibrillation who undergo percutaneous coronary intervention for coronary artery disease are treated with antiplatelet therapy on top of a non-vitamin K oral anticoagulant. Inevitably, this is associated with a higher risk of (major) bleeding. Given the reduction of ischemic risk with low-dose rivaroxaban and advances in stent properties, implantation techniques, and post-PCI management, it may be possible to treat atrial fibrillation patients after percutaneous coronary intervention with full-dose rivaroxaban and without antiplatelet therapy.

Objective: This study will serve as a pilot to investigate the feasibility and safety of rivaroxaban monotherapy in 50 patients with atrial fibrillation after percutaneous coronary intervention.

Study design: Single-centre, single arm pilot study with a stopping rule based on the occurrence of definite stent thrombosis Study population: Patients with atrial fibrillation and an indication for a non-vitamin K oral anticoagulant who undergo optimal percutaneous coronary intervention Intervention: Rivaroxaban 20 mg once daily or 15 mg once daily, in case of moderate-to-severe kidney dysfunction, for 6 or 12 months without antiplatelet therapy Main study endpoint: The primary ischemic endpoint is the composite of all-cause death, myocardial infarction, definite stent thrombosis, and ischemic stroke at 6 months after percutaneous coronary intervention. The primary bleeding endpoint is the composite of International Society on Thrombosis and Haemostasis defined major and clinically relevant non-major bleeding at 6 months after percutaneous coronary intevention.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Successful PCI
* History of or newly diagnosed (<72 hours after PCI/ACS) AF or atrial flutter with a long-term (≥ 1 year) indication for OAC
* Treatment with a loading dose of clopidogrel and aspirin prior to or during PCI

Exclusion Criteria:

* Known allergy or contraindication for rivaroxaban
* Current indication for OAC besides atrial fibrillation/flutter (e.g. venous thromboembolism)
* Overwriting indication for DAPT (e.g. TIA/CVA or PAD)
* Mechanical heart valve prosthesis
* Moderate to severe mitral valve stenosis (AVA ≤1.5 cm2)
* Intracardiac thrombus or apical aneurysm requiring OAC
* Kidney failure (eGFR <15)
* Active liver disease (ALT, ASP, AP >3x ULN or active hepatitis A, B or C)
* Active malignancy excluding non-melanoma skin cancer
* Active bleeding on randomization
* Severe anaemia requiring blood transfusion
* Pregnancy or breast-feeding women
* Planned high-bleeding risk surgical intervention within 6 months after PCI for stable CAD and 12 months after PCI for ACS
* PCI of left main disease, chronic total occlusion, bifurcation lesion requiring two-stent treatment, saphenous or arterial graft lesion, severely calcified lesions
* Participation in another trial with an investigational drug or device (i.e. stent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Primary ischemic endpoint | 6 months
  Composite of all-cause death, myocardial infarction, Academic Research Consortium defined definite stent trhombosis, or ischemic stroke
Primary bleeding endpoint | 6 months
  International Society on Thrombosis and Haemostasis defined major bleeding or clinically relevant non-major bleeding

IPD SHARING:
Plan to Share IPD: Undecided